CLINICAL TRIAL: NCT02878785
Title: Multicenter Phase 1/2 Study of Combination Therapy w/ DNA Methyltransferase Inhibitor Decitabine & Poly ADP Ribose Polymerase Inhibitor Talazoparib for Untreated AML in Adults Unfit for Cytotoxic Chemotherapy or R/R AML
Brief Title: Decitabine and Talazoparib in Untreated AML and R/R AML
Acronym: 1565GCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Pfizer (Industry); Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Maria Baer, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HP-00066370 1565GCC
Record Dates: First submitted 2016-08-03; First posted 2016-08-25 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1: Decitabine and Talazoparib Combo (Experimental): Phase 1:
  Decitabine by IV daily for 5 days every 28 days. Talazoparib orally daily days 1-28.
  The 'outer layer' of this nested dose escalation trial will escalate the dose of the two drugs by sequentially going through dose levels 1-6 in the table found in the protocol. The standard algorithm of the 3+3 design will be applied.
  Interventions: Drug: Decitabine; Drug: talazoparib
- Phase 2: Decitabine and Talazoparib Combo (Experimental): Phase 2:
  Recommended Phase 2 Dose (RP2D) The MTD of the combination of decitabine with a dose of talazoparib of at least 0.25 mg is defined as the maximal tolerated dose of decitabine studied - and for that dose level, combined with the maximum dose of talazoparib for which the incidence of DLT was less than 33% in 6 participants treated and this will be chosen as the recommended Phase 2 dose (RP2D). Among potential combined dose levels at MTD, available pharmacodynamic data (PARP trapping) will also be considered in the choice of RP2D, as will any significant indications of differences in clinical efficacy
  Interventions: Drug: Decitabine; Drug: talazoparib
- Phase 2 Arm A (Active Comparator): Adult patients with AML who are thought not to be likely to tolerate or respond to standard chemotherapy
  Interventions: Drug: Decitabine; Drug: talazoparib
- Phase 2 Arm B (Active Comparator): Adult patients with AML that has not responded to previous treatment or has come back after responding to previous treatment
  Interventions: Drug: Decitabine; Drug: talazoparib
- Phase 2 Arm C (Active Comparator): Adult patients previously treated with a DNA methyltransferase inhibitor (decitabine, azacitidine or guadecitabine)
  Interventions: Drug: Decitabine; Drug: talazoparib

INTERVENTIONS:
Drug: Decitabine — DNA methyltransferase inhibitor
  Other Names: dacogen
Drug: talazoparib — poly ADP ribose polymerase (PARP) inhibitor
  Other Names: BMN673; MDV3800

SUMMARY:
The purpose of this study is to find the best way to combine a new chemotherapy drug with one that is already in use to treat AML. The new experimental drug is called talazoparib (also known as BMN-673), and it is not approved by the Federal Drug Administration (FDA). The FDA is allowing the use of talazoparib for the purposes of this study.

Decitabine is used to treat bone marrow diseases called myelodysplastic syndromes (MDS), as well as off label for AML.

Lab work suggests that talazoparib will increase the effects of decitabine in leukemia cells.

Investigators hope that treating patients with decitabine and talazoparib together will be more successful that treating patients with decitabine alone.

This study has two parts. The purpose of part one the study is to find out the best doses of decitabine and talazoparib to use when they are given together to treat AML. The purpose of part two is to see how well the drugs work together to treat AML.

All participants in the study will be treated with decitabine and talazoparib.

Part one of the study will include as few as two people and as many as 36 people to find the best dose levels of the study drugs. Part one will begin enrolling first. Part two of the study will not start until the Part one of the study is complete. Participants will be told which part of the study they may be enrolled in. Part two of the study may include as few as 79 people and as many as 135 people. Part two includes three separate arms. Participants enrolled in Part two of the study, will be assigned to one of the three arms below in order to test the success rate of the study drug dose determined by Part one:

* Arm A will enroll adult patients with AML who are thought not to be likely to tolerate or respond to standard chemotherapy;
* Arm B will enroll adult patients with AML that has not responded to previous treatment or has come back after responding to previous treatment;
* Arm C will enroll adult patients previously treated with a DNA methyltransferase inhibitor (decitabine, azacitidine or guadecitabine).

This is a multi-center study. Up to 171 people may take part in this study globally.

DETAILED DESCRIPTION:
In this clinical trial, investigators combine decitabine and talazoparib in the treatment of patients with AML. Decitabine will be given in the established regimen of IV daily dosing for 5 days every 28 days. Talazoparib will be initiated orally daily on a continuous basis, beginning on Day 1 of Course 1. In this phase 1 trial, decitabine and talazoparib will be tested at 3 and 4 dose levels, respectively, yielding up to 6 combinations. Doses will be escalated based on tolerability using a 'classic' 3+3 design. Once the MTD for decitabine combined with 0.25 mg talazoparib is established, the dose of talazoparib will be escalated with the dose of decitabine kept fixed at the provisional MTD dose. There is no further stepping up or down of the drugs in the combination.

The regimen for phase 2 testing will be chosen based on tolerability, but also based on available pharmacodynamic and efficacy data. In phase 2, the selected combination regimen will be studied for efficacy.

Each patient will be treated until occurrence of either unacceptable toxicity or disease progression. Bone marrow aspirate and biopsy will be performed on approximately day 28 of each treatment course unless circulating blasts persist in the peripheral blood, until documentation of CR or CRi. Bone marrow aspirate and biopsy will then be repeated at time of clinical concern for disease progression.

In Phase 1, the clinical trial will enroll patients with relapsed and refractory AML in order to test the novel combination initially in patients with less favorable outcomes with decitabine alone. This is being done to avoid the possibility of compromising the outcomes of untreated patients, who have up to a 40% response rate to 5-day decitabine as a single agent, in the unlikely possibility that the combination is inferior. The regimen will then also be tested in previously untreated AML patients unfit for chemotherapy in phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML based on 2008 WHO criteria. AML may be de novo, following a prior hematologic disorder, including MDS or Philadelphia chromosome-negative myeloproliferative neoplasm, and/or therapy-related.
2. PHASES 1 AND 2: Patients with AML that has relapsed after, or is refractory to, first-line therapy, with or without subsequent additional therapy, and are currently considered unfit for, or unlikely to respond to, cytotoxic chemotherapy.
3. PHASE 2 ONLY: Patients previously untreated for AML who are considered unfit for cytotoxic chemotherapy by virtue of performance status, comorbidities, advanced age and/or low likelihood of response based on disease characteristics, or who decline cytotoxic induction chemotherapy.
4. Patients who have undergone autologous stem cell transplantation (autoSCT) are eligible provided that they are ≥ 4 weeks from stem cell infusion.
5. Patients who have undergone allogeneic SCT (alloSCT) are eligible if they are ≥ 60 days from stem cell infusion, have no evidence of graft versus host disease (GVHD) > Grade 1, and are ≥ 2 weeks off all immunosuppressive therapy.
6. Previous cytotoxic chemotherapy must have been completed at least 3 weeks and radiotherapy at least 2 weeks prior to Day 1 of treatment on the study, and all adverse events (excluding alopecia) due to agents administered more than 4 weeks earlier should have recovered to < Grade 1. Patients with hematologic malignancies are expected to have hematologic abnormalities at study entry. Hematologic abnormalities that are thought to be primarily related to leukemia are not considered to be toxicities (AE) and do not need to resolve to < Grade 1.
7. Prior DNA methyl transferase inhibitor administration (azacitidine, decitabine, or guadecitabine) for AML or for antecedent MDS is allowed if this clinical trial is considered the best treatment option, but azacitidine, decitabine, or guadecitabine must have been stopped at least 3 weeks prior to Day 1 of treatment on the study.
8. All biologic agents including hematopoietic growth factors must have been stopped at least 1 week prior to Day 1 of treatment on the study.
9. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of decitabine or talazoparib in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
10. ECOG performance status ≤2 (Karnofsky ≥60%).
11. Life expectancy of greater than 2 months.
12. Patients must have normal organ and marrow function as defined below:

    * Total bilirubin within normal institutional limits unless thought due to hemolysis or to Gilbert's syndrome;
    * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal;
    * Creatinine within normal institutional limits;

    OR

    • Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
13. Female patients of childbearing potential must have a negative pregnancy test, and female patients of childbearing potential and male patients must agree to use adequate contraception.

    Decitabine has been assigned to pregnancy category D by the FDA. Pregnant women must not take decitabine and female subjects must immediately stop taking decitabine and inform their doctor if they become pregnant during treatment. Decitabine is expected to result in adverse reproductive effects and can cause fetal harm when administered to a pregnant woman. In preclinical studies in mice and rats, decitabine was teratogenic, fetotoxic, and embryotoxic.

    Studies in pregnant animals to evaluate the effect of talazoparib on pregnancy have not been performed.

    Because decitabine is known to be teratogenic and the effects of talazoparib on the developing human fetus are unknown, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of decitabine and talazoparib administration.

    It is not known whether decitabine is excreted in human milk. Similarly, studies in lactating animals to evaluate the effect of talazoparib have not been performed, and thus, it is not known whether talazoparib is excreted in human milk. Therefore, breast-feeding should be stopped during decitabine and talazoparib treatment.
14. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia.
2. Patients with active central nervous system leukemia or requiring maintenance intrathecal chemotherapy.
3. Patients receiving concurrent chemotherapy, radiation therapy, or immunotherapy for AML.
4. Patients receiving any other investigational agents.
5. Hyperleukocytosis with >50,000 blasts/μl. Hydroxyurea for blast count control is permitted before starting treatment, but must be stopped prior to starting treatment on the study. Patients will be withdrawn from the study if > 50,000 blasts/μl occur or recur > 14 days after starting treatment on the study.
6. Active, uncontrolled infection. Patients with infection controlled with antibiotics are eligible.
7. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that per investigator's judgment would limit compliance with study requirements.
8. Patients who are pregnant or nursing.
9. Patients who have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks for antecedent malignancies prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or talazoparib.
11. Known HIV infection.

    HIV-positive patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
12. Previous treatment with talazoparib.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Baer, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Decitabine and Talazoparib Combo: Decitabine :10 mg/m^2: Period 1:: Participants were administered 10 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.25 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 8: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2: Period 1a:: Participants were administered 10 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.50 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 9: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2:: Participants were administered 15 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.25 mg of Talazopzrib orally diaily Days 1-28 at the same time each day
- Cohort 10: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2;Period 1b:: Participants were administered 10 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.75 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 11: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2;Period 1c:: Participants were administered 10 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 1.0 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 12: Decitabine and Talazoparib Combo:Decitabine :15 mg/m^2;Period 2a: Participants were administered 15 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.50 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 13: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2b:: Participants were administered 15 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.75 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 14: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2c:: Participants were administered 15 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 1.0 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 3: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 3:: Participants were administered 20 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.25 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 4: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 4:: Participants were administered 20 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.50 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 5: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 5:: Participants were administered 20 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 0.75 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 6: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 6:: Participants were administered 20 mg/m^2 of Decitabine intravenously (IV) daily for 5 days every 28 days. Participants were administered 1.0 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 7: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 7:: Participants were administered 20 mg/m^2 of Decitabine intravenously (IV) daily for 10 days every 28 days. Participants were administered 1.0 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
- Cohort 2:Decitabine 15 mg/m2 x 5 Days: Participants were administered 15 mg/m2 x 5 days every 28 days. Participants were administered .25 mg of Talazopzrib orally daily Days 1-28 at the same time each day.
Period: Overall Study
Arm/Group | Cohort 1: Decitabine and Talazoparib Combo: Decitabine :10 mg/m^2: Period 1: | Cohort 8: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2: Period 1a: | Cohort 9: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2: | Cohort 10: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2;Period 1b: | Cohort 11: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2;Period 1c: | Cohort 12: Decitabine and Talazoparib Combo:Decitabine :15 mg/m^2;Period 2a | Cohort 13: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2b: | Cohort 14: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2;Period 2c: | Cohort 3: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 3: | Cohort 4: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 4: | Cohort 5: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 5: | Cohort 6: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 6: | Cohort 7: Decitabine and Talazoparib Combo:Decitabine : 20 mg/m^2;Period 7: | Cohort 2:Decitabine 15 mg/m2 x 5 Days
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 3 | 3 | 3 | 3
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We completed the phase 1 study, but did not proceed to phase 2.
Groups:
- Phase 1: Decitabine and Talazoparib Combo: Phase 1:
  Decitabine by IV daily for 5 days every 28 days. Talazoparib orally daily days 1-28.
  The 'outer layer' of this nested dose escalation trial will escalate the dose of the two drugs by sequentially going through dose levels 1-6 in the table found in the protocol. The standard algorithm of the 3+3 design will be applied.
  Decitabine: DNA methyltransferase inhibitor
  talazoparib: poly ADP ribose polymerase (PARP) inhibitor
Arm/Group | Phase 1: Decitabine and Talazoparib Combo
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: The total overall enrollment was 25 patients. However, there were a total of 14 cohorts in this protocol and patients were enrolled over 7 of the 14 cohorts. Therefore, the analyzed patients in each row differs from the overall enrollment.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: <=18 years | 0
    Cohort 1: Between 18 and 65 years | 1
    Cohort 1: >=65 years | 2
    Cohort 2: number analyzed (Participants) | 3
    Cohort 2: <=18 years | 0
    Cohort 2: Between 18 and 65 years | 0
    Cohort 2: >=65 years | 3
    Cohort 3: number analyzed (Participants) | 3
    Cohort 3: <=18 years | 0
    Cohort 3: Between 18 and 65 years | 1
    Cohort 3: >=65 years | 2
    Cohort 4: number analyzed (Participants) | 7
    Cohort 4: <=18 years | 0
    Cohort 4: Between 18 and 65 years | 2
    Cohort 4: >=65 years | 5
    Cohort 5: number analyzed (Participants) | 3
    Cohort 5: <=18 years | 0
    Cohort 5: Between 18 and 65 years | 2
    Cohort 5: >=65 years | 1
    Cohort 6: number analyzed (Participants) | 3
    Cohort 6: <=18 years | 0
    Cohort 6: Between 18 and 65 years | 2
    Cohort 6: >=65 years | 1
    Cohort 7: number analyzed (Participants) | 3
    Cohort 7: <=18 years | 0
    Cohort 7: Between 18 and 65 years | 2
    Cohort 7: >=65 years | 1
    Cohort 8: number analyzed (Participants) | 0
    Cohort 8: <=18 years | 0
    Cohort 8: Between 18 and 65 years | 0
    Cohort 8: >=65 years | 0
    Cohort 9: number analyzed (Participants) | 0
    Cohort 9: <=18 years | 0
    Cohort 9: Between 18 and 65 years | 0
    Cohort 9: >=65 years | 0
    Cohort 10: number analyzed (Participants) | 0
    Cohort 10: <=18 years | 0
    Cohort 10: Between 18 and 65 years | 0
    Cohort 10: >=65 years | 0
    Cohort 11: number analyzed (Participants) | 0
    Cohort 11: <=18 years | 0
    Cohort 11: Between 18 and 65 years | 0
    Cohort 11: >=65 years | 0
    Cohort 12: number analyzed (Participants) | 0
    Cohort 12: <=18 years | 0
    Cohort 12: Between 18 and 65 years | 0
    Cohort 12: >=65 years | 0
    Cohort 13: number analyzed (Participants) | 0
    Cohort 13: <=18 years | 0
    Cohort 13: Between 18 and 65 years | 0
    Cohort 13: >=65 years | 0
    Cohort 14: number analyzed (Participants) | 0
    Cohort 14: <=18 years | 0
    Cohort 14: Between 18 and 65 years | 0
    Cohort 14: >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — Population: The total overall enrollment was 25 patients. However, there were a total of 14 cohorts in this protocol and patients were enrolled over 7 of the 14 cohorts. Therefore, the analyzed patients in each row differs from the overall enrollment.
  years
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1 | 75 [64 to 78]
    Cohort 2: number analyzed (Participants) | 3
    Cohort 2 | 75 [69 to 89]
    Cohort 3: number analyzed (Participants) | 3
    Cohort 3 | 69 [37 to 70]
    Cohort 4: number analyzed (Participants) | 7
    Cohort 4 | 73 [45 to 87]
    Cohort 5: number analyzed (Participants) | 3
    Cohort 5 | 63 [63 to 74]
    Cohort 6: number analyzed (Participants) | 3
    Cohort 6 | 57 [55 to 73]
    Cohort 7: number analyzed (Participants) | 3
    Cohort 7 | 55 [53 to 71]
    Cohort 8: number analyzed (Participants) | 0
    Cohort 9: number analyzed (Participants) | 0
    Cohort 10: number analyzed (Participants) | 0
    Cohort 11: number analyzed (Participants) | 0
    Cohort 12: number analyzed (Participants) | 0
    Cohort 13: number analyzed (Participants) | 0
    Cohort 14: number analyzed (Participants) | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total overall enrollment was 25 patients. However, there were a total of 14 cohorts in this protocol and patients were enrolled over 7 of the 14 cohorts. Therefore, the analyzed patients in each row differs from the overall enrollment.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: Female | 2
    Cohort 1: Male | 1
    Cohort 2: number analyzed (Participants) | 3
    Cohort 2: Female | 1
    Cohort 2: Male | 2
    Cohort 3: number analyzed (Participants) | 3
    Cohort 3: Female | 1
    Cohort 3: Male | 2
    Cohort 4: number analyzed (Participants) | 7
    Cohort 4: Female | 2
    Cohort 4: Male | 5
    Cohort 5: number analyzed (Participants) | 3
    Cohort 5: Female | 2
    Cohort 5: Male | 1
    Cohort 6: number analyzed (Participants) | 3
    Cohort 6: Female | 1
    Cohort 6: Male | 2
    Cohort 7: number analyzed (Participants) | 3
    Cohort 7: Female | 1
    Cohort 7: Male | 2
    Cohort 8: number analyzed (Participants) | 0
    Cohort 9: number analyzed (Participants) | 0
    Cohort 10: number analyzed (Participants) | 0
    Cohort 11: number analyzed (Participants) | 0
    Cohort 12: number analyzed (Participants) | 0
    Cohort 13: number analyzed (Participants) | 0
    Cohort 14: number analyzed (Participants) | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total overall enrollment was 25 patients. However, there were a total of 14 cohorts in this protocol and patients were enrolled over 7 of the 14 cohorts. Therefore, the analyzed patients in each row differs from the overall enrollment.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: Hispanic or Latino | 0
    Cohort 1: Not Hispanic or Latino | 3
    Cohort 1: Unknown or Not Reported | 0
    Cohort 2: number analyzed (Participants) | 3
    Cohort 2: Hispanic or Latino | 0
    Cohort 2: Not Hispanic or Latino | 3
    Cohort 2: Unknown or Not Reported | 0
    Cohort 3: number analyzed (Participants) | 3
    Cohort 3: Hispanic or Latino | 0
    Cohort 3: Not Hispanic or Latino | 3
    Cohort 3: Unknown or Not Reported | 0
    Cohort 4: number analyzed (Participants) | 7
    Cohort 4: Hispanic or Latino | 0
    Cohort 4: Not Hispanic or Latino | 7
    Cohort 4: Unknown or Not Reported | 0
    Cohort 5: number analyzed (Participants) | 3
    Cohort 5: Hispanic or Latino | 0
    Cohort 5: Not Hispanic or Latino | 3
    Cohort 5: Unknown or Not Reported | 0
    Cohort 6: number analyzed (Participants) | 3
    Cohort 6: Hispanic or Latino | 0
    Cohort 6: Not Hispanic or Latino | 3
    Cohort 6: Unknown or Not Reported | 0
    Cohort 7: number analyzed (Participants) | 3
    Cohort 7: Hispanic or Latino | 0
    Cohort 7: Not Hispanic or Latino | 3
    Cohort 7: Unknown or Not Reported | 0
    Cohort 8: number analyzed (Participants) | 0
    Cohort 9: number analyzed (Participants) | 0
    Cohort 10: number analyzed (Participants) | 0
    Cohort 11: number analyzed (Participants) | 0
    Cohort 12: number analyzed (Participants) | 0
    Cohort 13: number analyzed (Participants) | 0
    Cohort 14: number analyzed (Participants) | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The total overall enrollment was 25 patients. However, there were a total of 14 cohorts in this protocol and patients were enrolled over 7 of the 14 cohorts. Therefore, the analyzed patients in each row differs from the overall enrollment.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: American Indian or Alaska Native | 0
    Cohort 1: Asian | 0
    Cohort 1: Native Hawaiian or Other Pacific Islander | 0
    Cohort 1: Black or African American | 0
    Cohort 1: White | 3
    Cohort 1: More than one race | 0
    Cohort 1: Unknown or Not Reported | 0
    Cohort 2: number analyzed (Participants) | 3
    Cohort 2: American Indian or Alaska Native | 0
    Cohort 2: Asian | 0
    Cohort 2: Native Hawaiian or Other Pacific Islander | 0
    Cohort 2: Black or African American | 1
    Cohort 2: White | 2
    Cohort 2: More than one race | 0
    Cohort 2: Unknown or Not Reported | 0
    Cohort 3: number analyzed (Participants) | 3
    Cohort 3: American Indian or Alaska Native | 0
    Cohort 3: Asian | 0
    Cohort 3: Native Hawaiian or Other Pacific Islander | 0
    Cohort 3: Black or African American | 0
    Cohort 3: White | 3
    Cohort 3: More than one race | 0
    Cohort 3: Unknown or Not Reported | 0
    Cohort 4: number analyzed (Participants) | 7
    Cohort 4: American Indian or Alaska Native | 0
    Cohort 4: Asian | 1
    Cohort 4: Native Hawaiian or Other Pacific Islander | 0
    Cohort 4: Black or African American | 1
    Cohort 4: White | 5
    Cohort 4: More than one race | 0
    Cohort 4: Unknown or Not Reported | 0
    Cohort 5: number analyzed (Participants) | 3
    Cohort 5: American Indian or Alaska Native | 0
    Cohort 5: Asian | 0
    Cohort 5: Native Hawaiian or Other Pacific Islander | 0
    Cohort 5: Black or African American | 1
    Cohort 5: White | 2
    Cohort 5: More than one race | 0
    Cohort 5: Unknown or Not Reported | 0
    Cohort 6: number analyzed (Participants) | 3
    Cohort 6: American Indian or Alaska Native | 0
    Cohort 6: Asian | 0
    Cohort 6: Native Hawaiian or Other Pacific Islander | 0
    Cohort 6: Black or African American | 0
    Cohort 6: White | 3
    Cohort 6: More than one race | 0
    Cohort 6: Unknown or Not Reported | 0
    Cohort 7: number analyzed (Participants) | 3
    Cohort 7: American Indian or Alaska Native | 0
    Cohort 7: Asian | 0
    Cohort 7: Native Hawaiian or Other Pacific Islander | 0
    Cohort 7: Black or African American | 1
    Cohort 7: White | 2
    Cohort 7: More than one race | 0
    Cohort 7: Unknown or Not Reported | 0
    Cohort 8: number analyzed (Participants) | 0
    Cohort 9: number analyzed (Participants) | 0
    Cohort 10: number analyzed (Participants) | 0
    Cohort 11: number analyzed (Participants) | 0
    Cohort 12: number analyzed (Participants) | 0
    Cohort 13: number analyzed (Participants) | 0
    Cohort 14: number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Dose Finding
Description: To determine the recommended Phase 2 doses of Decitabine based on numbers of participants with treatment-related adverse events, evaluated according to Version 4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Cycle length = 28 days
Population: 25 patients with relapsed or refractory acute myeloid leukemia
Measure: Number; unit: mg/m^2
Groups:
- Cohort 1: Decitabine 10 mg/m^2 x 5 days Talazoparib 0.25 mg
- Cohort 2: Decitabine 15 mg/m^2 x 5 days Talazoparib 0.25 mg
- Cohort 3: Decitabine 20 mg/m^2 x 5 days Talazoparib 0.25 mg
- Cohort 4: Decitabine 20 mg/m^2 x 5 days Talazoparib 0.50 mg
- Cohort 5: Decitabine 20 mg/m^2 x 5 days Talazoparib 0.75 mg
- Cohort 6: Decitabine 20 mg/m^2 x 5 days Talazoparib 1.0 mg
- Cohort 7: Decitabine 20 mg/m^2 x 10 days Talazoparib 1.0 mg
- Cohort 8; Cohort 10; Cohort 11: Decitabine and Talazoparib Combo:Decitabine : 10 mg/m^2
- Cohort 9; Cohort 13; Cohort 14: Decitabine and Talazoparib Combo:Decitabine : 15 mg/m^2
- Cohort 12: Decitabine and Talazoparib Combo:Decitabine :15 mg/m^2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Cohort 13 | Cohort 14
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
mg/m^2 | 10 | 15 | 20 | 20 | 20 | 20 | 20 |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: After the subjects signed the consent until 30 days after the subjects finished treatment, an average of 1 year.
Description: Adverse Events were not collected/monitored individually for each dose level. Arms/Groups were combined when reporting AEs and SAEs per PI discretion as only the overall toxicity data was collected and submitted and published in a medical journal.
Groups:
- Phase 1 Dose Escalation: Decitabine in combination with Talazoparib
Arm/Group | Phase 1 Dose Escalation
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 25/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (N=25)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 8 (25)
Infection (Respiratory, thoracic and mediastinal disorders) | 15 (25) — Infection, lung
Sepsis/bacteremia (Infections and infestations) | 12 (25)
Fungal infection (Infections and infestations) | 2 (25)
Other infections (Infections and infestations) | 8 (25)
Fever (Infections and infestations) | 19 (25)
Intracranial bleed (Nervous system disorders) | 2 (25)
Pericardial tamponade (Cardiac disorders) | 1 (25)
Atrial fibrillation (Cardiac disorders) | 3 (25)
Vomiting (Gastrointestinal disorders) | 1 (25)
Diarrhea (Gastrointestinal disorders) | 2 (25)
Transaminitis (Hepatobiliary disorders) | 1 (25)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (25)
Elevated creatinine (Renal and urinary disorders) | 1 (25)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation (N=25)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Other infections (Infections and infestations) | 1 (1)
Other infections (Infections and infestations) | 5 (5)
Fever (Immune system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Transaminitis (Hepatobiliary disorders) | 3 (3)
Elevated creatinine (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT02878785/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT02878785/ICF_001.pdf